CLINICAL TRIAL: NCT03862521
Title: Safety of Low and Very Low Carbohydrate Diets in Young Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LowCHOT1D
Record Dates: First submitted 2019-02-26; First posted 2019-03-05 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes Mellitus; Diet Modification; Child, Only
Keywords: type 1 diabetes; low carbohydrate diets; insulin pump therapy; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: randomized to either low or very low carbohydrate diet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carbohydrate diet group (Experimental): Low carb diet, carbohydrates make up 30-40% of total daily calories.
  Interventions: Other: Low carbohydrate diet
- Very low carbohydrate diet (Experimental): Very low carb diet, carbohydrates make up 20-29% of total daily calories.
  Interventions: Other: Very low carbohydrate diet

INTERVENTIONS:
Other: Low carbohydrate diet — Low carbohydrate diet
  Arms: Low carbohydrate diet group
Other: Very low carbohydrate diet — Very low carbohydrate diet
  Arms: Very low carbohydrate diet

SUMMARY:
The purpose of the study is to evaluate the safety of short-term (6 month) low or very-low carbohydrate diets in prepubertal children 2 to <12 years old with type 1 diabetes. Participants will be randomized to either low carbohydrate diet (carbohydrate makes up 30-39% of total daily calories) or very-low carbohydrate diet (carbohydrates are 20-29% of total daily calories). The investigators will evaluate metabolic effects of these diets by measuring the counter-regulatory hormone response to hypoglycemia at baseline and again at 3 months. Other outcomes include diabetes control as measured by HbA1c, growth and weight gain, lipid profiles, and body composition.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety of short-term (6 month) low or very-low carbohydrate diets in prepubertal children 2 to <12 years old with type 1 diabetes. Participants will be randomized to either low carbohydrate diet (carbohydrate makes up 30-39% of total daily calories) or very-low carbohydrate diet (carbohydrates are 20-29% of total daily calories). The investigators will evaluate metabolic effects of these diets by measuring the counter-regulatory hormone response to hypoglycemia at baseline and again at 3 months. Other outcomes include diabetes control as measured by HbA1c, growth and weight gain, lipid profiles, and body composition.

Participants will be admitted to the Clinical Research Center at baseline and 3 months. Gradual reduction in serum glucose to under 80 mg/dL will be achieved by an increase in their insulin infusion rate through their insulin pump. Plasma glucose, catecholamines (epinephrine, norepinephrine), glucagon, and serum ketones are measured at baseline and after glucose is below 80 mg/dL. All subjects will have lipid evaluation and body composition (DXA scan) at baseline and 6 months. Subjects' growth will be evaluated by comparing their height and weight z-score before and after the 6 months of diet intervention. Change in growth velocity will also be assessed. During the study, participants not already using continuous glucose monitoring will be placed on Dexcom G5 to monitor blood sugars regularly. Subjects will also be monitoring serum ketones at home regularly.

ELIGIBILITY:
Inclusion criteria

* Prepubertal children 2 to <12 years old (i.e., before 12th birthday)
* Type 1 diabetes for at least 6 months
* Patients must be using insulin pump therapy
* Not presently on low carbohydrate diet

Exclusion criteria

* On low or very low carbohydrate diet
* History of endocrine or metabolic disorder that could affect counter-regulation (well-controlled hypothyroidism is acceptable if on stable dose of l-thyroxine for ≥3 months)
* History of metabolic disorder affection lipid metabolism
* Severe hypoglycemic event in past 3 months

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in hormone (epinephrine, norepinephrine, glucagon) response to hypoglycemia | Baseline to 3 months
  Change from baseline to 3 months in the hormone (epinephrine, norepinephrine, glucagon) response to insulin-induced hypoglycemia.

SECONDARY OUTCOMES:
Change in height in centimeters from baseline to 6 months | Baseline to 6 months
  Change in height in centimeters from baseline to 6 months
Change in weight in kilograms from baseline to 6 months | Baseline to 6 months
  Change in weight in kilograms from baseline to 6 months
Change in body composition from baseline to 6 months | Baseline to 6 months
  Change in percent body fat using DXA scan from baseline to 6 months
Change in A1c from baseline to 3 and 6 months | Change from baseline to 3 and 6 months
  Change in A1c over the length of the study
Change in lipid profile from baseline to 6 months | Baseline to 6 months
  Change in lipid profile from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Fox, MD, Principal Investigator — Nemours Children's Health
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No